CLINICAL TRIAL: NCT05696236
Title: Transepidermal Water Loss as a Predictor for Severe Allergic Reactions in Oral Food Challenges
Brief Title: Predicting Peanut Anaphylaxis and Reducing Epinephrine
Acronym: PrePARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Principal Investigator, Charles (Chase) Schuler, Assistant Professor of Allergy and Clinical Immunology and Assistant Professor of Mary H Weiser Food Allergy, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: HUM00205852
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Anaphylaxis Food
Keywords: Allergic reaction to food; Water loss across the skin; Food challenge
MeSH Terms: interventions — Monitoring, Physiologic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants and families, the food allergy nurse administering the oral food challenge (OFC), and the allergist physician assessing and treating the patient will be blinded to the study arm status.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Monitor (TEWL) and stopping rules (Experimental): Wears the monitor, and the food challenge will be done using the new stopping rules to end the test.
  Interventions: Device: Transepidermal water loss (TEWL) monitor and stopping rules
- Monitor (TWLG) without stopping rules (Active Comparator): Wears the monitor, but the stopping rules will not be used to end the food challenge. The food challenge will be done following standard oral food challenge procedures.
  Interventions: Device: Monitor (TEWL) without stopping rules

INTERVENTIONS:
Device: Transepidermal water loss (TEWL) monitor and stopping rules — The oral food challenge will be done as usual, and participants will wear the TEWL monitor. The research food allergy nurse and doctor will also be looking for signs and symptoms of an allergic reaction. The research study coordinator will be watching the TEWL numbers. If they numbers match the stopping rules, they will tell the doctor and the oral food challenge will be over.
  Arms: Monitor (TEWL) and stopping rules
Device: Monitor (TEWL) without stopping rules — The oral food challenge will be done as usual, and participants will wear the TEWL monitor. The research food allergy nurse and doctor will be looking for signs and symptoms of an allergic reaction. The research study coordinator will be watching the TEWL numbers, but the stopping rules will not be used to end the oral food challenge.
  Arms: Monitor (TWLG) without stopping rules

SUMMARY:
This research study is testing a new way to look for the early stages of anaphylaxis. Eligible participants will have a small monitor (transepidermal water loss) placed on the forearm during a food challenge (for peanut allergies). This monitor continuously records the amount of water lost through the skin.

In a previous study the team learned what values are associated with an anaphylactic reaction. These values are called "stopping rules." This study is looking at whether it can use these new stopping rules to end the oral food challenge before a person may show any symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Have a known history of food anaphylaxis to peanut confirmed by an allergist
* Have had skin and blood food allergy testing to peanut within the past 12 months. Meet the 80% likelihood positive predictive value threshold for peanut allergy based on at least 1 of either the skin or blood immunoglobulin E (IgE) tests per current literature corrected for age.
* Meet all clinical oral food challenge (OFC) requirements. This includes no asthma or atopic dermatitis exacerbations, no recent viral infections, no recent antibiotics, and no food allergy reactions in the past month.

Exclusion Criteria:

* Any known cardiovascular disease, cancer, pulmonary disease except well-controlled asthma, or other condition that would preclude an OFC otherwise.
* Any medication use that would interfere with an OFC result. Medications in this category include antihistamines (first or second generation) within 1 week, omalizumab within 3 months, and others listed in the protocol appendix.
* Any skin condition aside from well-controlled eczema that might impact TEWL measurement, including such conditions as autoimmune skin conditions (such as psoriasis), congenital ichthyoses, hyper-IgE syndromes.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chase Schuler, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Freigeh GE, O'Shea KM, Troost JP, Kaul B, Franco LM, Schuler CF 4th. Transepidermal Water Loss in Oral Food Challenges in Children With Peanut Allergy: A Randomized Clinical Trial. JAMA Netw Open. 2025 Nov 3;8(11):e2543371. doi: 10.1001/jamanetworkopen.2025.43371. PMID 41236740

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to randomization, 3 participants were screen fails and 2 were lost to follow up.
Period: Overall Study
Arm/Group | Monitor (TEWL) and Stopping Rules | Monitor (TWLG) Without Stopping Rules
Started | 21 | 25
Completed | 18 | 22
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Later determined to not be eligible for participation | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monitor (TEWL) and Stopping Rules | Monitor (TWLG) Without Stopping Rules | Total
Number analyzed (Participants) | 21 | 25 | 46
Age, Continuous [Mean (Standard Deviation); unit: months] | 34 (17.2) | 29 (14.3) | 31 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 14 | 13 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 21 | 23 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 18 | 23 | 41
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 25 | 46

OUTCOME MEASURES:

1. Primary Outcome: Anaphylaxis Occurrence Rates in Each Group
Description: Any Brighton Level 1, 2, or 3 anaphylaxis. The Brighton Level is a system for classifying the severity and diagnostic certainty of anaphylaxis cases, particularly in the context of adverse events following immunization. Results reflect the number of participants who experienced any of the Brighton Level 1, 2, or 3 anaphylaxis events.
Time Frame: Approximately 4-6 hours (Day 1 during the food challenge)
Population: 6 participants ended their participation in the trial before their data was collectible.
Measure: Count of Participants; unit: Participants
Arm/Group | Monitor (TEWL) and Stopping Rules | Monitor (TWLG) Without Stopping Rules
Number analyzed (Participants) | 18 | 22
Participants | 9 | 10
Statistical Analysis 1: Comparison: Monitor (TEWL) and Stopping Rules vs Monitor (TWLG) Without Stopping Rules; Test type: Superiority; p = 0.77, t-test, 2 sided

2. Secondary Outcome: Reaction Rates in Each Group
Description: Results reflect the number of participants who experienced any objective symptom of allergic reaction (e.g., hives, angioedema, vomiting, wheeze, etc) not rising to the definition of anaphylaxis.
Time Frame: Approximately 4-6 hours (Day 1 during the food challenge)
Population: 6 participants ended their participation in the trial before their data was collectible.
Measure: Count of Participants; unit: Participants
Arm/Group | Monitor (TEWL) and Stopping Rules | Monitor (TWLG) Without Stopping Rules
Number analyzed (Participants) | 18 | 22
Participants | 16 | 14
Statistical Analysis 1: Comparison: Monitor (TEWL) and Stopping Rules vs Monitor (TWLG) Without Stopping Rules; Test type: Superiority; p = 0.07, t-test, 2 sided

3. Secondary Outcome: Anaphylaxis Severity in Each Group
Description: Anaphylaxis severity was graded on a scale of 1 to 5 (where 1 = mild, 5 = death)) according to criteria set forth in the Consortium for Food Allergy Research (CoFAR) Grading Scale.
Time Frame: Approximately 4-6 hours (Day 1 during the food challenge)
Population: 6 participants ended their participation in the trial before their data was collectible.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Monitor (TEWL) and Stopping Rules | Monitor (TWLG) Without Stopping Rules
Number analyzed (Participants) | 18 | 22
score on a scale | 1.8 (0.75) | 2.6 (0.51)
Statistical Analysis 1: Comparison: Monitor (TEWL) and Stopping Rules vs Monitor (TWLG) Without Stopping Rules; Test type: Superiority; p = 0.006, t-test, 2 sided

4. Secondary Outcome: Anaphylaxis Likelihood in Each Group Based on the Brighton Score
Description: The Brighton score was a 1-3 score of anaphylaxis likelihood. Participants were categorized based on level of anaphylaxis likelihood: Not Applicable (no reaction), Brighton Level 1 (most likely), Brighton Level 2 (medium likelihood), Brighton Level 3 (least likely), Unclassified (reaction present, but with insufficient symptoms for participant's reaction to be classified)
Time Frame: Approximately 4-6 hours (Day 1 during the food challenge)
Population: 6 participants ended their participation in the trial before their data was collectible.
Measure: Count of Participants; unit: Participants
Arm/Group | Monitor (TEWL) and Stopping Rules | Monitor (TWLG) Without Stopping Rules
Number analyzed (Participants) | 18 | 22
Participants
  Not Applicable | 3 | 8
  Brighton Level 1 | 3 | 2
  Brighton Level 2 | 4 | 7
  Brighton Level 3 | 2 | 1
  Unclassified | 6 | 4

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Monitor (TEWL) and Stopping Rules | Monitor (TWLG) Without Stopping Rules
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 16/18 | 14/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monitor (TEWL) and Stopping Rules (N=18) | Monitor (TWLG) Without Stopping Rules (N=22)
Allergic Reaction (Immune system disorders) | 16 | 14 — All reactions were food allergy reactions up to food anaphylaxis. There is no single definition for food anaphylaxis, so all food-reaction adverse events are reported here.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT05696236/Prot_SAP_000.pdf